CLINICAL TRIAL: NCT06474117
Title: Muscle-tendon Interaction in the Spastic Sural Triceps During Gait
Acronym: GEcho
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: Laboratoire Motricité, Interactions, Performance (MIP) (Unknown); Société Française de Physiothérapie (SFP). (Unknown)
Responsible Party: Sponsor
Other Study IDs: RC24_0274; 2024-A01157-40 (Other: ANSM (IDRCB))
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-06

CONDITIONS: Spinal Cord Injuries; Stroke
Keywords: Gait; Echography; Spinal Cord Injury; Stroke
MeSH Terms: conditions — Spinal Cord Injuries; Stroke | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Post-Stroke Patients: Patients will undergo gait analysis coupled with ultrasound to measure the lengths of the Achilles tendon and gastrocnemius medialis muscle. They will also have their force/length profile of the GM measured on an isokinetic dynamometer with simultaneous ultrasound
  Interventions: Other: Gait analysis coupled with ultrasound; Other: Isokinetic dynamometer with simultaneous ultrasound
- Post-Spinal Cord Injury Patients: Similar to the post-stroke group, these patients will undergo gait analysis coupled with ultrasound to measure the lengths of the Achilles tendon and gastrocnemius medialis muscle. The force/length profile of the GM will also be measured on an isokinetic dynamometer with simultaneous ultrasound.
  Interventions: Other: Gait analysis coupled with ultrasound; Other: Isokinetic dynamometer with simultaneous ultrasound
- Healthy controls: The healthy control group will undergo the same gait analysis and ultrasound measurements as the patient groups. Their force/length profile of the GM will also be measured on an isokinetic dynamometer with simultaneous ultrasound for comparison with the post-stroke and post-spinal cord injury groups.
  Interventions: Other: Gait analysis coupled with ultrasound; Other: Isokinetic dynamometer with simultaneous ultrasound

INTERVENTIONS:
Other: Gait analysis coupled with ultrasound — Measure the lengths of the Achilles tendon and gastrocnemius medialis muscle
Other: Isokinetic dynamometer with simultaneous ultrasound — Measure the force/length profile of the gastrocnemius medialis muscle

SUMMARY:
This project aims to study the mechanical behavior of the muscle-tendon unit (MTU) of the gastrocnemius medialis (GM) and the Achilles tendon (AT) in post-stroke and spinal cord injured (SCI) patients compared to a healthy population, focusing on the variations in muscle and tendon length during the stance phase of the gait cycle. The primary objective is to assess the respective contributions of the GM and AT lengthening in the MTU during walking. Inclusion criteria include adult post-stroke and post-SCI patients with voluntary motor function and some walking capacity. Methods include ultrasound measurements and 3D gait analysis.

DETAILED DESCRIPTION:
Primary Objective: Evaluate the respective contributions of the gastrocnemius medialis (GM) muscle and the Achilles tendon (AT) within the muscle-tendon unit (MTU) during the single support phase of walking in post-stroke patients compared to healthy subjects.

Study Description: Strokes often lead to spastic paresis, degrading patients' walking performance. Instrumented gait analysis allows for the evaluation of these performances to propose adapted therapeutic strategies. This project will compare muscle and tendon behavior during walking between healthy individuals and post-stroke patients.

Methodology:

* Participants: Adult post-stroke patients or incomplete SCI patients with voluntary motor function on the triceps surae and walking capacity. Control group composed of healthy adults.
* Procedures:

  * Measure the force/length profile of the GM on an isokinetic dynamometer with simultaneous ultrasound.
  * Conduct gait analysis coupled with ultrasound to measure the lengths of the AT and GM.
  * Compare muscle and tendon length data during the stance phase of the gait cycle between the two groups.

ELIGIBILITY:
Inclusion Criteria :

Post-Stroke Population:

* Adult male or female
* Patient who had a stroke more than 7 days ago
* Patient hospitalized (in conventional hospitalization or day hospital) in the university neurological rehabilitation department of CHU de Nantes
* Patient with voluntary motor function graded between 2 and 4 on the MRC (Medical Research Council) scale at the GM level
* Patient classified between 3 and 8 on the New Functional Ambulation Classification

Post-Spinal Cord Injury Population:

* Adult male or female
* Patient with an incomplete spinal cord injury classified as ASIA AIS C or D from level C2 to L5
* Patient hospitalized (in conventional hospitalization or day hospital) in the neurological rehabilitation department of CHU de Nantes
* Patient with voluntary motor function graded between 2 and 4 on the MRC (Medical Research Council) scale at the GM level
* Patient classified between 3 and 8 on the New Functional Ambulation Classification

Healthy Population:

• Adult male or female without any neurological disorders

Exclusion Criteria :

Post-Stroke and Post-Spinal Cord Injury Population:

* Minor patient
* History of calf surgery, surgery to reduce triceps surae spasticity, or intramuscular injection (e.g., botulinum toxin) in the plantar flexors within the last 6 months
* Patient with a progressive condition contraindicating physical exertion (e.g., syrinx, cardiovascular instability)
* Peripheral pathology of the considered lower limb

Healthy Population:

* History of calf surgery
* History of muscle injury, fracture, or sprain of the lower limb within the last 3 months
* History of neurological disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects, post-stroke subject, SCI subjects
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2026-11-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Length of the Achilles Tendon (AT), Muscle Fibers of the Gastrocnemius Medialis (GM), and the Muscle GM During the Single Support Phase of Walking | 1 Day
  This measure involves the use of ultrasound to assess the lengths of the Achilles tendon, muscle fibers of the gastrocnemius medialis, and the entire muscle GM during the single support phase of the gait cycle in post-stroke and SCI patients compared to healthy controls. The primary goal is to determine the contributions of the muscle and tendon to the overall muscle-tendon unit during walking.

SECONDARY OUTCOMES:
Positioning of the Muscle Fibers on the Force-Length Curve During Different Phases of Walking | 1 Day
  This outcome measure evaluates the positioning of the muscle fibers of the gastrocnemius medialis on the force-length curve during various phases of the gait cycle, including the single support phase and the double support phases (reception and propulsion). The measurements will be compared between post-stroke, SCI patients and healthy controls. The assessment will involve ultrasound measurements and isokinetic dynamometry to determine the force-length relationship.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nantes, Nantes, Loire Atlantique, France

IPD SHARING:
Plan to Share IPD: No